CLINICAL TRIAL: NCT01930773
Title: Optimal P2Y12-receptor treatmeNt Guided by bedSIDe Genetic or Pharmacodynamic TESTing to Prevent Periprocedural Myonecrosis During Elective Percutaneous Coronary Intervention.
Brief Title: Bedside Genetic or Pharmacodynamic Testing to Prevent Periprocedural Myonecrosis During PCI (ONSIDE TEST)
Acronym: ONSIDE TEST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Polish Cardiac Society (Other); University of Pecs (Other)
Responsible Party: Principal Investigator, Łukasz Kołtowski, Cardiology Researcher, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONSIDE TEST; Klub 30, 2012 (Other: Polish Cardiac Society)
Record Dates: First submitted 2013-08-25; First posted 2013-08-29 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Stable Angina
Keywords: clopidogrel; prasugrel; platelet function testing; genotyping; peri-procedural MI
MeSH Terms: conditions — Angina, Stable | interventions — Genotyping Techniques; Immunophenotyping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Genotyping Arm (Experimental): Rapid genotyping to select optimal P2Y12-inhibitor for PCI.
  Interventions: Device: Genotyping
- Phenotying Arm (Experimental): The use of platelet function testing to select the optimal P2Y12-inhibitor for PCI.
  Interventions: Device: Phenotyping
- Conventional Arm (No Intervention): Regular approach for performing elective PCI.

INTERVENTIONS:
Device: Genotyping — Patients harboring CYP2C19 *2 alleles receive 60 mg prasugrel for PCI, while non-carriers receive 600 mg clopidogrel if not pretreated with clopidogrel.
  Other Names: Spartan rapid genotyping device to screen CYP2C19 *2 carriage in patients in the Genotyping Arm.
  Arms: Genotyping Arm
Device: Phenotyping — Patients having high on-treatment platelet reactivity (HPR: greater than 208 PRU) receive 60 mg prasugrel loading dose (LD), others continue clopidogrel for PCI.
  Other Names: VerifyNow P2Y12 assay to test the response to clopidogrel.
  Arms: Phenotying Arm

SUMMARY:
Patients undergoing percutaneous coronary intervention with a residual high platelet reactivity despite oral clopidogrel are at increased risk of ischaemic complications. The strategies to overcome the issue consist of switch to a more potent antiplatelet medications including prasugrel or ticagrelor. Economic constrains of many countries still do not allow wide reimbursement of newer antiplatelet agents. Therefore a strategy to personalise treatment according to genotype and phenotype characteristics of the patient may provide an attractive solution combining high clinical efficacy with low budget impact.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* elective PCI

Exclusion Criteria:

* acute coronary syndrome (troponin > 1 x ULN),
* administration of glycoprotein IIb/IIIa inhibitors,
* chronic total occlusion,
* lesions with extensive calcifications requiring rotational atherectomy,
* platelet count <70 000 /µl
* high bleeding risk,
* coronary bypass surgery in the previous 3 months,
* severe chronic renal failure (eGFR < 30 mL/min)
* requirement for warfarin, dabigatran, apixaban, rivaroxaban
* history of stroke or TIA,
* weight < 60 kg
* known bleeding diathesis,
* hematocrit of < 30% or >52%
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of periprocedural myocardial injury within 24 h after PCI | Within 24 hours after Percutaneous Coronary Intervention (PCI)
  Post-procedural troponin value increase exceeding the 99th percentile upper reference limit (URL) within 24 hours after PCI

SECONDARY OUTCOMES:
Proportion of patients having periprocedural myocardial infarction (MI) | Within 24 hours or PCI
  Periprocedural MI is defined as a CK-MB elevation greater than 3x of the upper limit of norm (ULN) within 24 hours of elective PCI.

OTHER OUTCOMES:
Peak troponin elevation | Within 24 hours of PCI
  The level of peak troponin-I elevation during 24 hours of elective PCI
Proportion of patients with peri-procedural MI | Within 24 hours of PCI
  The rate of peri-procedural MI defined as a peak troponin-I value greater than 5x the ULN within 24 hours.
BARC type 3 and 5 bleeding | Within 1 week of PCI
  BARC-defined type 3 (clinical, laboratory, and/or imaging evidence of bleeding, with healthcare provider responses) and type 5 (fatal) bleeds happening within 7 days of PCI.
Death, MI, stent thrombosis (ST) or urgent repeat revascularization | 30 days after PCI
  The rate of cardiac death, myocardial infarction, definite or probable stent thrombosis or urgent repeat revascularization within 30 days of elective PCI.

CONTACTS AND LOCATIONS:
Locations (2):
- Heart Center Balatonfüred, Balatonfüred, Hungary
- 1st Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Koltowski L, Aradi D, Huczek Z, Tomaniak M, Sibbing D, Filipiak KJ, Kochman J, Balsam P, Opolski G. Study design and rationale for Optimal aNtiplatelet pharmacotherapy guided by bedSIDE genetic or functional TESTing in elective percutaneous coronary intervention patients (ONSIDE TEST): a prospective, open-label, randomised parallel-group multicentre trial (NCT01930773). Kardiol Pol. 2016;74(4):372-9. doi: 10.5603/KP.a2015.0172. Epub 2015 Sep 14. PMID 26365936
- Available data/document: Study Protocol — http://www.ncbi.nlm.nih.gov/pubmed/26365936 — Study design and rationale for Optimal aNtiplatelet pharmacotherapy guided by bedSIDE genetic or functional TESTing in elective percutaneous coronary intervention patients (ONSIDE TEST): a prospective, open-label, randomised parallel-group multicentre trial (NCT01930773). Kołtowski Ł, Aradi D, Huczek Z, Tomaniak M, Sibbing D, Filipiak KJ, Kochman J, Balsam P, Opolski G. Kardiol Pol. 2016;74(4):372-9. doi: 10.5603/KP.a2015.0172.
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/28281736 — Optimal aNtiplatelet pharmacotherapy guided by bedSIDE genetic or functional TESTing in elective PCI patients: A pilot study: ONSIDE TEST pilot. Koltowski L, Tomaniak M, Aradi D, Huczek Z, Filipiak KJ, Kochman J, Gajda S, Balsam P, Opolski G. Cardiol J. 2017 Mar 10. doi: 10.5603/CJ.a2017.0026. [Epub ahead of print]